CLINICAL TRIAL: NCT02206529
Title: Enhancing Family Based Treatment of Childhood Obesity Through Social Networks
Acronym: CONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 211098
Record Dates: First submitted 2014-07-21; First posted 2014-08-01 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Child Obesity
Keywords: obesity; child; weight management; behavioral; social networks; social support
MeSH Terms: conditions — Pediatric Obesity; Obesity; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Social Network Engagement+Std Treatment (Active Comparator): Social Network Engagement = content and activities to help the parent engage his/her social network in supporting healthy lifestyle behaviors.
  Standard Treatment = family-based behavioral pediatric obesity treatment, as per protocol outlined in FOCUS trial (Family Overweight: Comparing Use of Strategies; NCT00746629)
  Interventions: Behavioral: Social Network Engagement+Std Treatment
- Standard Treatment (Other): This comparator arm consists of historical controls, participants in the FOCUS trial who received standard treatment.
  Standard Treatment = family-based behavioral pediatric obesity treatment, as per protocol outlined in FOCUS trial (Family Overweight: Comparing Use of Strategies; NCT00746629)
  Interventions: Behavioral: Standard Treatment

INTERVENTIONS:
Behavioral: Social Network Engagement+Std Treatment
  Other Names: SNE
  Arms: Social Network Engagement+Std Treatment
Behavioral: Standard Treatment — Standard Treatment = family-based behavioral pediatric obesity treatment, as per protocol outlined in FOCUS trial (Family Overweight: Comparing Use of Strategies; NCT00746629)
  Other Names: FOCUS Intervention
  Arms: Standard Treatment

SUMMARY:
The purpose of this study is to develop a Social Network Engagement (SNE) Intervention that will be integrated into a standard treatment program for childhood overweight. The investigators will conduct a pilot trial of SNE to assess feasibility and to estimate its effectiveness compared with historical controls who received standard treatment. The historical controls will be participants in the FOCUS trial (Family Overweight: Comparing Use of Strategies; NCT00746629).

ELIGIBILITY:
Inclusion Criteria Children

* Age 7-13 years
* At or above the 85th percentile for age- and gender-specific BMI

Parents

• At least one overweight parent (BMI>25.0)

Parents and children

* English-speaking and at least at a second-grade reading level
* Live <50 miles from the treatment site.

Exclusion Children

* Conditions known to promote obesity (e.g., Prader-Willi),
* Participation in another weight control program
* Recently started taking weight-affecting medications (e.g., stimulants).

Parents and children

* Disability or illness that would preclude them from engaging in at least moderate-intensity physical activity,
* Current or prior diagnosed eating disturbance
* Thought disorder, suicidality, or substance abuse disorder

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Child BMI Z-score | 20 weeks after baseline
Child BMI Z-score | One year post-treatment

SECONDARY OUTCOMES:
Peds QL (child self-report and parent report) | 20 weeks after baseline
  Pediatric Quality of Life Score
Parent BMI | 20 weeks after baseline
  Intervention is aimed at the parent-child dyad, so parent weight status is assessed.
Peds QL (child self-report and parent report) | One year post-treatment
  Pediatric Quality of Life Score
Parent BMI | One year post-treatment
  Intervention is aimed at the parent-child dyad, so parent weight status is assessed.

OTHER OUTCOMES:
SSQ (Social Support Questionnaire-Short Form) | 20 weeks after baseline
  Global social support measure, assessed as possible mediator of effect of intervention on primary and secondary outcomes.
QRI (Quality of the Relationship Index) | 20 weeks after baseline
  Relationship-specific social support measure, assessed as possible mediator of effect of intervention on primary and secondary outcomes.
SPSI-R (Social Problem-Solving Index-for Research) | 20 weeks after baseline
  Measure of parental skill in problem-solving, assessed as possible mediator of effect of intervention on primary and secondary outcomes.
Behavioral Skill Assessment | 20 weeks after baseline
  Process measure of parental use of skills taught during intervention
WMSI (Weight Management Support Index) | 20 weeks after baseline
  Measure of parental perceived social support related to weight management, assessed as possible mediator of primary and secondary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Lozano, MD MPH, Principal Investigator — Group Health Research Institute